CLINICAL TRIAL: NCT04107753
Title: The Impact of Brief Motivational Counseling for Smoking Cessation in an Italian Emergency Department: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Collaborators: Lega Italiana per la Lotta contro i Tumori (Other)
Responsible Party: Principal Investigator, Fabrizio Faggiano, Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CE 93/16
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Smoking Habit
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Patients in whom the inclusion criteria are met are asked by the triage nurses if they are smokers. Those patients are then asked by the triage nurses if they want to participate in the study; those who consent are randomized in the control or intervention group. The triage window of the software currently used for clinical care management in the ED (PsNet, Hi. Tech Spa) has been equiped in such a way that, for patients who agree to participate in the study, is casually print one of the two symbols on the informative consent paper given to patient in the end of the triage procedure.
Who Masked: Participant
Masking Description: Patients do not know in which group they were randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Brief counseling based on the 5As model (Experimental): The intervention group received a brief counseling based on the 5As model. It mainly consists of the following steps: ask, advice, asses, assist, arrange. It is performed by the nurse who take clinical care of the patient. The patients receive an information card about the Smoke cessation center's (CTT) and the patients who agree are contacted by the CTT's staff.
  Interventions: Behavioral: Brief counseling based on the 5As model
- Control group (No Intervention): No other intervention than the "usual care" (range between the not mentioning the subject at all, to a general advice to quit without bringing any evidence or any structured counseling).

INTERVENTIONS:
Behavioral: Brief counseling based on the 5As model — It is a structured brief counselling perfomed by nurse who takes clinical care of the patient and it is performed as follow:
  1. ASK: every patient should be asked whether he/she is or is not a smoker;
  2. ADVICE: the patient is advised to quit in a strong, clear and personalized way;
  3. ASSESS: the patient is asked if he/she would like to quit and the strenght of his/her dependence is assessed.
  4. ASSIST: The smoker interested in quitting are assisted in their attempts, for example by helping them to define a quit date, by advising them about strategies against withdrawal symptoms and by providing them information material; patients are asked whether they want to be contacted by the CTT.
  5. ARRANGE: this step is only addressed to the patients who have started a treatment in the CTT and is expected to prevent or treat eventual relapses.
  Arms: Intervention: Brief counseling based on the 5As model

SUMMARY:
Smoke is still a significant Public Health problem. The Emergency Departments (EDs) could be the ideal setting to set up smoke cessation interventions (high prevalence of smoking patient compared to the general population). The structured brief counseling 5As based (ask, advice, asses, assist, arrange) is an effective Public Health intervention when performed by the General Practitioners. Still not clear is its feasibility and effectiveness in the ED setting. Aim of the study. To assess the feasibility and effectiveness of the 5As based counselling in the University ED of Novara compared to the "usual care".

DETAILED DESCRIPTION:
The study is a Randomized Controlled Trial performed in Novara (Piedmont, Italy) in the ED of the "Maggiore della Carità" University Hospital and involving the Treatment Center for Tobacco use (CTT) of the Addiction Department of the Local Health Unit of Novara (ASL NO).

The RCT has two parallel groups (allocation 1:1): the intervention group and the controll group.

Adult smokers attending ED of the "Maggiore della Carità" University Hospital of the city of Novara are invited to participate to the intervention.

The intervention consists in the "5As" smoke cessation brief structured counselling performed by the ED nurses. The 5As counselling is composed by 5 main steps:

1. Ask: every patient is asked whether he/she is or is not a smoker in order to identify those who could benefit from the counseling;
2. Advice: the patient is advised to quit in a strong, clear and personalized way;
3. Assess: the patient is asked if he/she would like to quit and it is assessed the strength of his/her dependence in order to tailor the following step on the patient's situation and readiness to quit;
4. Assist: all the patients receive the counseling by the nurse and those interested in quitting are assisted in their attempts. Furthermore patients are asked whether they want to be contacted by the CTT in order to start an intensive treatment;
5. Arrange: for the patients willing to make a quit attempt, it is aimed to arrange for follow up contact by the CTT and to start a treatment in the CTT. It is expected also to prevent or treat eventual relapses.

The controll group received no intervention ("usual care" that could range between not mentioning the subject at all, to a general advice to quit without bringing any structured counselling).

All the nurses involved in the project as "intervention providers" will receive a proper training carried out by the CTT staff. The training will be focused on:

* the description and application of the 5As intervention;
* the importance of the relationship with patients;
* the acquisition of specific skills through role playing techniques.

The sample size needed is 1200 patients (600 for each arm of the study). This sample size has been calculated assuming that:

* in Italy the annual cessation rate in the general population is 8.4% (Istituto Superiore di Sanità, 2015);
* that the relative risk of 12-month point-estimated tobacco abstinence in the intervention group compared to the general population is 1.6.

The calculation was based on desired significance level of 5% (two-tailed) and power of 80%.

The evaluation of the feasibility and sustainability of the intervention is descriptive and the investigators did not include it in the power calculation.

Data collection. Data about patients are collected as follow:

* through the ED software; the ED software records all the clinically relevant information (triage, visit, observation and monitoring, if needed, or discharge);
* from the baseline questionnaire. Patients from both groups will be given a questionnaire about their smoking habits in order to collect data about their health status, socio-demographic characteristics, their degree of addiction by using the Fagerström test and their orientation with respect to the possibility of quitting. The questionnaire is the adaptation of the already validated questionnaire of the FRITT project, implemented in Sweden from the Karolinska Institutet, with the addition of the Fageström test for nicotine dependence. It also takes inspiration from the questionnaire SPRINT.
* from the nurse checklist. The check list is filled by the nurses involved in the study at the moment of the contact with the patients of the intervention group. The check list is aimed to investigate if the intervention has been carried out and in detail which steps have been performed. In the event that the intervention had not been carried out, the reason for this is collected in the check list;
* from the follow up- questionnaire. The follow-up questionnaire is administered by telephone at 6 and 12 month in order to collect the informations about the outcomes. Participants in the follow-up phase will be contacted by telephone at least 3 times at different hours of the day, in order to maximize the possibilities to get an answer.
* from the CTT software for those who decided to proceed with the intensive treatment.

All the data collected are recorded in the Research Electronic Data Capture (RedCap). RedCap is a secure web application that ensures the confidentiality of the data and high privacy levels, according to the Italian law.

Results will be analyzed with "intention-to treat" principle: each patient will be considered under original randomization no matter what counseling he/she actually received. In secondary analyzes, the investigators will perform both "per protocol" and "as treated" analyses.

Data monitoring. Due to the short duration of the trial and to the lack of recognized collateral effects, there is no need of a data monitoring committee.

The project does not implicate any physical intrusion or risk for participants.

Consent or assent is obtained first orally by the triage nurse than written by a designated person.

Access to data. The only actors who will have access to the final trial dataset are the researchers of Eastern Piedmont University involved in the study and the CTT physicians who collaborated at the study.

ELIGIBILITY:
Inclusion Criteria:

* self-statement as "current smokers" (at least one cigarette per day) during the triage interview;
* age ≥ 18;
* priority code urgency (yellow code) or deferrable urgency (green code) or non-urgency (white code);
* provision of an informed consent.

Exclusion Criteria:

* priority code emergency (red code);
* altered mental status or history of psychiatric illness;
* inability to understand either written or oral Italian;
* patient already in treatment or follow-up for tobacco addiction;
* patient allocated to a nurse who has not been trained in counseling and does not participate to the study;
* informed consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
Point prevalence of tobacco-free patients assessment | At 12 months from the intervention
  Those who did not smoke in the last 7 days; dichotomous variable: yes/no. Better outcome: yes. Investigated by the ad-hoc telephone administrated questionnaire.

SECONDARY OUTCOMES:
Point prevalence of tobacco-free patients assessment | At 6 months from the intervention
  Those who did not smoke in the last 7 days; dichotomous variable: yes/no. Better outcome: yes.
  Investigated by the ad-hoc telephone administrated questionnaire.
Continuous abstinence during the last 3 months assessment | At 12 months from the intervention
  Categorical variable treated as a dichotomous one (yes/no). Better outcome: yes. Investigated by the ad-hoc telephone administrated questionnaire.
Decrease of at least 50% in daily tobacco use in the past 7 days with respect to baseline | At 12 months from the intervention
  Continuous variable categorized in a dichotomous one:
  has there been a 50% decrease in daily tobacco use in the past 7 days with respect to baseline? Yes/no. Better outcome: yes. Variable used as a dichotomous one for the statistical analysis. Investigated by the ad-hoc telephone administrated questionnaire.
Transition in motivational stages | At 12 months from the intervention
  The follow stages of the Transtheoretical Model of behavior change were investigated by the ad-hoc telephone administrated questionnaire: precontemplation, preparation, action and maintenance stages. The categoric variable is used as a dichotomous one: has the transition from one stage of change to another occurred? Yes/no. The outcome is positive when the passage from one stage of change to another towards the direction of the maintenance stage occurs.
Quit attempts number. | At 12 months from the intervention
  Continuous variable used as dichotomous one: has there been at least one quit attempt (including cessation) in the last six month occurred? Yes/no. Investigated by the ad-hoc telephone administrative questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi del Piemonte Orientale "Amedeo Avogadro", Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foulds J. Strategies for smoking cessation. Br Med Bull. 1996 Jan;52(1):157-73. doi: 10.1093/oxfordjournals.bmb.a011523. PMID 8746304
- [Background] Gorini G, Carreras G, Giordano L, Anghinoni E, Iossa A, Coppo A, Talassi F, Galavotti M, Chellini E; SPRINT Working Group. The Pap smear screening as an occasion for smoking cessation and physical activity counselling: effectiveness of the SPRINT randomized controlled trial. BMC Public Health. 2012 Sep 5;12:740. doi: 10.1186/1471-2458-12-740. PMID 22950883
- [Background] Lancaster T, Stead LF. Individual behavioural counselling for smoking cessation. Cochrane Database Syst Rev. 2002;(3):CD001292. doi: 10.1002/14651858.CD001292. PMID 12137623
- [Background] McBride CM, Emmons KM, Lipkus IM. Understanding the potential of teachable moments: the case of smoking cessation. Health Educ Res. 2003 Apr;18(2):156-70. doi: 10.1093/her/18.2.156. PMID 12729175
- [Background] Patrick DL, Cheadle A, Thompson DC, Diehr P, Koepsell T, Kinne S. The validity of self-reported smoking: a review and meta-analysis. Am J Public Health. 1994 Jul;84(7):1086-93. doi: 10.2105/ajph.84.7.1086. PMID 8017530
- [Background] Virtanen SE, Zeebari Z, Rohyo I, Galanti MR. Evaluation of a brief counseling for tobacco cessation in dental clinics among Swedish smokers and snus users. A cluster randomized controlled trial (the FRITT study). Prev Med. 2015 Jan;70:26-32. doi: 10.1016/j.ypmed.2014.11.005. Epub 2014 Nov 18. PMID 25445335